CLINICAL TRIAL: NCT06415643
Title: The Use of Islet Organoids in the Treatment of Pancreatic Surgery-related Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Newislet Biotechnology (Shanghai) Ltd. (Unknown)
Responsible Party: Principal Investigator, Sheng Yan, Professor, MD, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YD-ZE-001
Record Dates: First submitted 2024-05-09; First posted 2024-05-16 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: T3c Diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transplantation group (Experimental): transplantation group
  Interventions: Other: Islet organoids transplantation

INTERVENTIONS:
Other: Islet organoids transplantation — autologous transplantation of ex vivo expanded islet organoids.

SUMMARY:
The purpose of this clinical trial is to verify the safety and effectiveness of autologous islet organoids transplantation after in vitro expansion for the treatment of pancreatogenic diabetes.

DETAILED DESCRIPTION:
The purpose of this clinical trial is to verify the safety and effectiveness of autologous islet transplantation after in vitro expansion in the forms of functional islet organoids, for the treatment of pancreatogenic diabetes in participants who have undergone pancreatic resection through a single-center single-arm study. The investigators aim to establish the entire operational process of isolating expanding and transplanting islets from the pancreas removed from the participants and managing postoperative care. The investigators hope to accumulate clinical experience in treating pancreatogenic diabetes with transplanted autologous islet cell clusters expanded in vitro establish standard and regulated medical operations and gather materials for future applications of this treatment method in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form and adhere to the trial treatment plan and visit schedule.
2. When signing the informed consent form, the age should be between 18-70 years old, with no gender restrictions.
3. Good overall health condition: no damage to important organs such as heart, lungs, liver, kidneys, no serious or uncontrolled infections, and no history of severe mental disorders.
4. Meets the diagnosis of pancreatic tumor, chronic pancreatitis (diffuse pancreatic duct stones, refractory pain, associated with high risk of pancreatic cancer), pancreatic trauma, postoperative pancreatic fistula with class C, pancreatic cystic fibrosis, has indications for total or subtotal pancreatectomy, and no chronic organ failure.
5. Clinical examinations must meet the following criteria: Normal glycated hemoglobin (HbA1c) measurement.
6. Normal alanine aminotransferase (ALT) measurement, or abnormal but clinically insignificant
7. negative for Hepatitis A virus antibody (HAV antibody), Hepatitis B virus surface antigen (HBsAg) and e antigen, Hepatitis C virus antibody (HCV antibody), Human Immunodeficiency Virus antibody (HIV-1 and HIV-2 antibody), Syphilis antibody, Epstein-Barr virus antibody (EBV antibody), Cytomegalovirus (CMV-DNA), B19 virus nucleic acid, Human T-lymphotropic virus antibody.
8. Male participants who are sexually active and have not undergone surgical sterilization or whose partners are capable of childbearing, agree to take effective contraceptive measures for the entire trial period and at least 6 months after the end of the study, and not to donate sperm. Female participants capable of childbearing agree to take effective contraceptive measures for the entire study period and at least 6 months after the end of the study.
9. Post-pancreatic surgery blood sugar increase, meeting the diagnostic criteria for diabetes (World Health Organization 2019 edition).
10. C-peptide level <0.3 ng/mL 120 minutes after mixed meal stimulation before pancreatic islet transplantation.

Exclusion Criteria:

1. The investigator considers the following diseases to be clinically significant: a history of diabetes, or preoperative hyperglycemia, meeting the diagnosis of diabetes.
2. Undergone previous pancreatic or islet transplantation
3. Uncontrolled hypertension, such as systolic blood pressure (SBP) >160 mmHg and/or diastolic blood pressure (DBP) >100 mmHg after treatment with a stable dose (at least 4 weeks) of antihypertensive drugs.
4. Fatty hepatitis, portal vein thrombosis, portal hypertension, anterolateral pancreatic jejunostomy, or visceral hyperalgesia.Impaired liver and kidney function at screening (reference to the normal range of laboratory tests in the research center): aspartate aminotransferase (AST) >3 times the upper limit of normal (ULN), alanine aminotransferase (ALT) >3 times ULN, total bilirubin level (TBL) >2 times ULN (excluding Gilbert's syndrome). Creatinine clearance <45 mL/min (calculated by Cockcroft-Gault formula)
5. Women in pregnancy, less than 6 months after miscarriage, less than 1 year after delivery and lactation.
6. History of infectious diseases including but not limited to hepatitis A, hepatitis B, hepatitis C, HIV and syphilis
7. Presence of known hemoglobin-related diseases, anemia (moderate to severe) or other known hemoglobin diseases that interfere with HbA1c measurement (such as sickle cell disease). Presence of massive albuminuria (urinary protein excretion rate >300 mg/g) or past medical history.
8. Presence of severe heart disease or cardiovascular disease within 6 months before screening, including: stroke, decompensated heart failure (NYHA class III or IV), myocardial infarction, unstable angina, those who have undergone coronary artery bypass grafting.
9. History of coagulation disorders or need for long-term anticoagulation treatment (such as warfarin) (low-dose aspirin treatment is allowed) or INR>1.5
10. Treatment (local, intra-articular, intraocular, or inhaled formulations) for any other factors or diseases, other than the above reasons, that the researcher deems unsuitable for participation in this clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-08-10 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
C-peptide secretion | before transplantation and 1 year after transplantation
  C-peptide detection assay

SECONDARY OUTCOMES:
HbA1c level | before transplantation and 1 year after transplantation
  HbA1c detection assay
Mean Amplitude of Glycemic Excursion (MAGE) | 12 weeks and 52 weeks post transplantation
  Glucose measurement
Ryan Hypoglycemia event | baseline and 52 weeks post transplantation
  recorded events of unaware severe hypoglycemia (glucose level below 3 mmol/L)
Reduced Insulin usage | 12 weeks and 52 weeks post transplantation
  Reduced insulin usage of over 50% compared with prior to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Yan, PhD, MD, Principal Investigator — Zhejiang University Second Affiliated Hospital
Locations (1):
- Zhejiang University Second Affiliated Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No